CLINICAL TRIAL: NCT03092375
Title: A Phase 3b, Multi-Center, Randomized, Open-Label, Pragmatic Study of Glecaprevir/Pibrentasvir (G/P) +/- Ribavirin for GT1 Subjects With Chronic Hepatitis C Previously Treated With an NS5A Inhibitor + Sofosbuvir Therapy
Brief Title: Multi-Center, Randomized, Open-Label Study of G/P +/- RBV for NS5A + SOF Previously Treated GT1 HCV Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B16-439; OCR16260 (Other: University of Florida)
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Hepatitis C; HCV
Keywords: HCV; Previously treated
MeSH Terms: conditions — Hepatitis C | interventions — glecaprevir; pibrentasvir; glecaprevir and pibrentasvir; Ribavirin; Tablets

STUDY DESIGN:
Intervention Model Description: Main Study Up to 225 subjects will be enrolled into 4 study arms A, B, C and D with Glecaprevir/Pibrentasvir (G/P) with or without Ribavirin (RBV).
  About 75-90 non-cirrhotic subjects will be randomized in a 2:1 ratio to Arms A and B, and about 110-135 compensated cirrhotic subjects will be randomized in a 1:1 ratio to Arms C and D.
  Non-cirrhotic subjects will be randomized 2:1 to:
  1. Arm A: G/P 300 mg/120 mg Once a day for 12 weeks
  2. Arm B: G/P 300 mg/120mg Once a day for 16 weeks
     Subjects with compensated cirrhosis will be randomized 1:1 to:
  3. Arm C: G/P 300 mg/120 mg QD + weight-based RBV (Ribavirin) Twice a day (1000 mg or 1200 mg total daily dose) for 12 weeks
  4. Arm D: G/P 300 mg/120 mg QD for 16 weeks Retreatment sub-study Up to 11 subjects who still have hepatitis C virus after being treated in the Main study will have the option to enter the Retreatment sub-study and receive G/P plus Sofosbuvir and with or without RBV.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A: G/P 300 mg/120 mg QD for 12 Wks (Experimental): Non-cirrhotic subjects will take Glecaprevir/Pibrentasvir (G/P) 300mg/120mg (3 Glecaprevir/Pibrentasvir (G/P) 100mg/40mg Tablets once-daily by mouth) for 12 weeks.
  Interventions: Drug: Glecaprevir/Pibrentasvir (G/P) 300mg/120mg
- Arm B: G/P 300 mg/120 mg QD for 16 Wks (Experimental): Non-cirrhotic subjects will take Glecaprevir/Pibrentasvir (G/P) 300mg/120mg once-daily by mouth for 16 weeks (G/P 300 mg/120 mg QD for 16 Wks)
  Interventions: Drug: Glecaprevir/Pibrentasvir (G/P) 300mg/120mg
- Arm C: G/P 300 mg/120 mg QD + RBV 12 Wks (Experimental): Cirrhotic subjects will take Glecaprevir/Pibrentasvir (G/P) 300mg/120mg once daily plus Ribavirin 200Mg Tablet (2-3 tablets) twice a day for 12 weeks (G/P 300 mg/120 mg QD + RBV 12 Wks)
  Interventions: Drug: Glecaprevir/Pibrentasvir (G/P) 300mg/120mg; Drug: Ribavirin 200Mg Tablet
- Arm D: G/P 300 mg/120 mg QD for 16 Wks (Experimental): Cirrhotic subjects will take Glecaprevir/Pibrentasvir (G/P) 300mg/120mg once daily for 16 weeks (G/P 300 mg/120mg QD for 16 Wks)
  Interventions: Drug: Glecaprevir/Pibrentasvir (G/P) 300mg/120mg

INTERVENTIONS:
Drug: Glecaprevir/Pibrentasvir (G/P) 300mg/120mg — daily
  Other Names: Glecaprevir/Pibrentasvir; GLE/PIB (Glecaprevir/Pibrentasvir)
Drug: Ribavirin 200Mg Tablet — Weight-based 1000-1200 mg
  Other Names: Ribasphere 200Mg Tablet
  Arms: Arm C: G/P 300 mg/120 mg QD + RBV 12 Wks

SUMMARY:
The study will enroll well-compensated cirrhotic as well as non-cirrhotic subjects treatment experienced with an NS5a Inhibitor + sofosbuvir and will include patients who did not complete the prescribed duration due to adverse event or any reason other than for non/poor compliance. Subjects will be randomized to 12 or 16 weeks of treatment.

DETAILED DESCRIPTION:
The primary purpose of this study is to compare the efficacy and safety of glecaprevir and pibrentasvir (G/P) for 12 weeks to G/P for 16 weeks in non-cirrhotic NS5A (non-structural protein 5a)-inhibitor plus sofosbuvir ± RBV (Ribavirin) treatment-experienced adults with HCV genotype 1 (GT1) infection, and to compare the efficacy and safety of G/P with RBV for 12 weeks to G/P without RBV for 16 weeks in NS5A-inhibitor plus sofosbuvir (SOF) ± RBV treatment-experienced adults with compensated cirrhosis and GT1 infection.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 18 years of age at time of screening.
2. A history of previous treatment with an NS5A-inhibitor plus sofosbuvir therapy ± RBV for chronic HCV genotype 1 infection.
3. Treatment must have been completed at least 1 month prior to Screening Visit.
4. Screening laboratory result indicating chronic HCV GT1 infection. Subjects must be able to understand and adhere to the study visit schedule and all other protocol requirements and must voluntarily sign and date an informed consent.

Exclusion Criteria:

1. History of severe, life-threatening or other significant sensitivity to any drug.
2. Female who is pregnant, planning to become pregnant during the study or breastfeeding; or male whose partner is pregnant or planning to become pregnant during the study.
3. Recent (within 6 months prior to study drug administration) history of drug or alcohol abuse that could preclude adherence to the protocol in the opinion of the investigator.
4. Positive test result at Screening for hepatitis B surface antigen (HBsAg) or anti-human immunodeficiency virus antibody (HIV Ab) in patient without known history of HIV infection.
5. HCV genotype performed during screening indicating co-infection with more than one HCV genotype.
6. History or presence of liver decompensation.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2020-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Nelson, MD, Principal Investigator — University of Florida
Locations (31):
- United States (31):
  - Stanford University, Palo Alto, California
  - University of California, San Francisco, San Francisco, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Health Research Institute, Washington D.C., District of Columbia
  - UF Hepatology Research at CTRB, Gainesville, Florida
  - UF Health Jacksonville-Gastroenterology Emerson, Jacksonville, Florida
  - Schiff Center for Liver Diseases/University of Miami, Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Atlanta Medical Center, Atlanta, Georgia
  - Atlanta Gastro Associates, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - The Johns Hopkins Hospital/John G. Bartlett Specialty Practice, Baltimore, Maryland
  - Digestive Disease Associates, PA, Catonsville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Univ. of Minnesota Health Clinics and Surgery Center, Inc., Minneapolis, Minnesota
  - Southern Therapy and Advanced Research, Jackson, Mississippi
  - Northwell Health - Sandra Atlaas Bass Center for Liver Diseases, Manhasset, New York
  - NYU Langone Medical Center, New York, New York
  - Weill Cornell Medicine, Hepatology, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - University of Pennsylvania-Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Bon Secours Liver Institute of Virginia, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang GP, Schnell GL, Kort JJ, Sidhu GS, Schuster L, Tripathi RL, Larsen L, Michael LC, Bergquist K, Magee A, Patel CB, Whitlock JA, Tamashiro R, Peter JA, Fried MW, Nelson DR. Linkage of resistance-associated substitutions in GT1 sofosbuvir + NS5A inhibitor failures treated with glecaprevir/pibrentasvir. J Hepatol. 2021 Oct;75(4):820-828. doi: 10.1016/j.jhep.2021.04.057. Epub 2021 May 21. PMID 34023351
- [Derived] Lok AS, Sulkowski MS, Kort JJ, Willner I, Reddy KR, Shiffman ML, Hassan MA, Pearlman BL, Hinestrosa F, Jacobson IM, Morelli G, Peter JA, Vainorius M, Michael LC, Fried MW, Wang GP, Lu W, Larsen L, Nelson DR. Efficacy of Glecaprevir and Pibrentasvir in Patients With Genotype 1 Hepatitis C Virus Infection With Treatment Failure After NS5A Inhibitor Plus Sofosbuvir Therapy. Gastroenterology. 2019 Dec;157(6):1506-1517.e1. doi: 10.1053/j.gastro.2019.08.008. Epub 2019 Aug 8. PMID 31401140

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A: G/P 300 mg/120 mg QD for 12 Wks | Arm B: G/P 300 mg/120 mg QD for 16 Wks | Arm C: G/P 300 mg/120 mg QD + RBV 12 Wks | Arm D: G/P 300 mg/120 mg QD for 16 Wks
Started | 78 | 49 | 21 | 29
Completed | 78 | 48 | 20 | 29
Not Completed | 0 | 1 | 1 | 0
Not completed — Lack of Efficacy | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: G/P 300 mg/120 mg QD for 12 Wks | Arm B: G/P 300 mg/120 mg QD for 16 Wks | Arm C: G/P 300 mg/120 mg QD + RBV 12 Wks | Arm D: G/P 300 mg/120 mg QD for 16 Wks | Total
Number analyzed (Participants) | 78 | 49 | 21 | 29 | 177
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 53 | 31 | 16 | 16 | 116
  >=65 years | 25 | 18 | 5 | 13 | 61
Age, Continuous [Mean (Full Range); unit: years] | 60.99 [40 to 77] | 61.37 [45 to 75] | 59.10 [38 to 70] | 62.59 [42 to 81] | 61.3 [38 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 5 | 6 | 34
  Male | 64 | 40 | 16 | 23 | 143
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 32 | 25 | 8 | 12 | 77
  White | 44 | 23 | 12 | 17 | 96
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 1 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 78 | 49 | 21 | 29 | 180
HCV Genotype, non-1b [Count of Participants; unit: Participants] — HCV Genotype was characterized as 1b and non-1b
  Participants | 60 | 39 | 17 | 26 | 142
HCV RNA [Median (Full Range); unit: LOG10 IU/mL] — Baseline HCV RNA, log10 IU/ML, MEDIAN (RANGE)
  LOG10 IU/mL | 6.4 [1.9 to 7.7] | 6.4 [4.0 to 7.7] | 6.3 [5.1 to 7.0] | 6.4 [3.7 to 7.1] | 6.4 [1.9 to 7.7]
PLATELET [Median (Full Range); unit: 10E3 cells/uL] — Platelets collected at Baseline Lab Draw
  10E3 cells/uL | 204.50 [30 to 370] | 193 [100 to 343] | 125 [46 to 270] | 134 [63 to 253] | 178 [30 to 370]
ALT [Median (Full Range); unit: u/L] | 41 [11 to 611] | 38 [13 to 208] | 59 [33 to 171] | 70 [23 to 166] | 45 [11 to 611]
APRI [Median (Full Range); unit: Index] — AST to Platelet Ratio Index (APRI) (AST Level (IU/L)/AST (Upper Limit of Normal) (IU/L))/Platelet Count (109/L) * 100
  Index | .46 [.11 to 6.06] | .45 [.17 to 2.39] | 1.23 [.41 to 6.58] | 1.47 [.24 to 3.37] | .57 [.11 to 6.58]
Estimated GFR [Median (Full Range); unit: ml/min/1.73M2] — Estimated Glomerular Filtration Rate
  ml/min/1.73M2 | 88.36 [27.36 to 136.70] | 86.08 [42.94 to 134.53] | 94.99 [75.23 to 138.27] | 96.61 [60.34 to 167.09] | 90.41 [27.36 to 167.09]
HIV [Count of Participants; unit: Participants] — Number of patients with HIV at baseline
  Participants | 5 | 2 | 1 | 1 | 9
Albumin [Median (Full Range); unit: g/dL] | 4.10 [3.20 to 4.70] | 4.10 [2.90 to 4.60] | 4.10 [3.20 to 4.50] | 3.90 [3.20 to 4.50] | 4.10 [2.90 to 4.70]

OUTCOME MEASURES:

1. Primary Outcome: SVR After G/P 12 Wks (Arm A) vs. G/P Given for 16 Weeks (Arm B) to Non-cirrhotic Treatment-experienced GT1 HCV Participants
Description: Number of non-cirrhotic treatment-experienced HCV genotype 1 with a NS5Ai inhibitor + SOF +/-RBV participants with undetectable HCV RNA (HCV RNA <Lower Limit of Quantification -LLOQ) 12 weeks after completing G/P 300 mg/100 mg daily for 12 weeks (Arm A) vs. 16 weeks of G/P 300 mg/100 mg daily (Arm B)
Time Frame: Up to 28 weeks
Population: These analyses were completed on Modified ITT -Genotype Population defined as all treated subjects representing their actual study regimen and who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: G/P 300 mg/120 mg QD for 12 Wks | Arm B: G/P 300 mg/120 mg QD for 16 Wks
Number analyzed (Participants) | 78 | 49
Participants
  Virologic Response | 70 | 46
  Virologic Failure | 8 | 3

2. Primary Outcome: Comparison of Cirrhotic Participants Achieving SVR 12 After G/P Plus RBV for 12 Wks vs. G/P for 16 Wks
Description: Number of cirrhotic participants who are treatment experienced with a NS5A inhibitor + SOF +/RBV with undetectable HCV RNA 12 weeks after completing G/P plus RBV for 12 wks vs. G/P for 16 Wks
Time Frame: Up to 28 weeks
Population: Cirrhotic subjects achieving Virologic Response at Post-Treatment Week 12
Measure: Count of Participants; unit: Participants
Groups:
- Arm D: G/P 300 mg/120 mg QD for 16 Wks: Arm D includes Cirrhotic subjects receiving Glecaprevir/Pibrentasvir (G/P) 300mg/120mg once daily for 16 weeks (G/P 300 mg/120mg QD for 16 Wks)
  Glecaprevir/Pibrentasvir (G/P) 300mg/120mg: daily
Arm/Group | Arm C: G/P 300 mg/120 mg QD + RBV 12 Wks | Arm D: G/P 300 mg/120 mg QD for 16 Wks
Number analyzed (Participants) | 21 | 29
Participants
  Virologic Response | 18 | 28
  Virologic Failure | 3 | 1

3. Primary Outcome: Tolerability of G/P +/-RBV
Description: Number of subjects who discontinued G/P due to adverse events
Time Frame: Up to 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: G/P 300 mg/120 mg QD for 12 Wks | Arm B: G/P 300 mg/120 mg QD for 16 Wks | Arm C: G/P 300 mg/120 mg QD + RBV 12 Wks | Arm D: G/P 300 mg/120 mg QD for 16 Wks
Number analyzed (Participants) | 78 | 49 | 21 | 29
Participants | 0 | 0 | 0 | 0

4. Secondary Outcome: Difference in On-Treatment Virologic Failure Between Arms A & B (Non-cirrhotic Subjects)
Description: Difference in % of subjects with on-treatment virologic failure further defined as either 1)Breakthrough a)Confirmed HCV RNA ≥ 100 IU/mL after HCV RNA < Lower Limit of Quantification (LLOQ) at some point during the Treatment Period or confirmed increase from nadir in HCV RNA (two consecutive measurements > 1 log10 IU/mL above nadir) at any time point during the Treatment Period, or b) a single value indicating viral breakthrough (≥ 100 IU/mL or > 1 log10 above nadir), followed by patient status of 'Lost to Follow-up', the latter not requiring confirmation by a proximate measurement) or 2) End of Treatment Failure defined as HCV RNA ≥ LLOQ at end of treatment and following at least 6 weeks of treatment.
Time Frame: Up to 28 weeks
Population: Analysis was performed the study population "as treated" further defined as mITT-all subjects representing their actual study regimen and who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Arms A G/P 300 mg/120 mg QD for 12 Weeks: Arms A includes non-cirrhotic subjects receiving Glecaprevir/Pibrentasvir (G/P) 300mg/120mg once-daily by mouth with or without Ribavirin for 12 weeks (Arm A) Glecaprevir/Pibrentasvir (G/P) 300mg/120mg: daily
- Arm B G/P 300/120mg Once Daily for 16 Weeks: Arm B includes non-cirrhotic subjects receiving Glecaprevir/Pibrentasvir (G/P) 300mg/120mg once-daily by mouth for 16 weeks (G/P 300 mg/120 mg QD for 16 Wks)
  Glecaprevir/Pibrentasvir (G/P) 300mg/120mg: daily
Arm/Group | Arms A G/P 300 mg/120 mg QD for 12 Weeks | Arm B G/P 300/120mg Once Daily for 16 Weeks
Number analyzed (Participants) | 78 | 49
Participants | 1 | 1
Statistical Analysis 1: Comparison: Arms A G/P 300 mg/120 mg QD for 12 Weeks vs Arm B G/P 300/120mg Once Daily for 16 Weeks; The difference in the percentage of subjects with on-treatment virologic failure (Defined as increase of >1 log10 IU/mL above nadir during treatment, or HCV RNA >= 15 IU/mL at end of treatment with at least 6 weeks of treatment between Arms A and B are summarized with two-sided 95% Wilson score intervals; Test type: Other — Study is not intended to be powered; Mean Difference (Final Values) = -0.76, 95% CI 2-sided [-9.48 to 5.12] — Excludes re-infection and death

5. Secondary Outcome: Difference in Relapse Between Arms A & B in Non-cirrhotic Subjects
Description: Difference in Post-treatment relapse (defined as confirmed HCV RNA>= Lower limit of quantification (LLOQ) between end of treatment and 12 weeks after the last dose of study drug among subjects who completed treatment as planned with HCV RNA < LLOQ at end of treatment, excluding subjects with subjects with reinfection)
Time Frame: Up to 28 weeks
Population: Analysis performed on any subject with study drug duration of 77 days or greater for Arm A or 105 days or greater for Arm B
Measure: Count of Participants; unit: Participants
Groups:
- Arm A: G/P 300 mg/120 mg QD for 12 Wks: Non-cirrhotic subjects receiving Glecaprevir/Pibrentasvir (G/P) 300mg/120mg (3 Glecaprevir/Pibrentasvir (G/P) 100mg/40mg Tablets once-daily by mouth) for 12 weeks.
  Glecaprevir/Pibrentasvir (G/P) 300mg/120mg: daily
Arm/Group | Arm A: G/P 300 mg/120 mg QD for 12 Wks | Arm B: G/P 300 mg/120 mg QD for 16 Wks
Number analyzed (Participants) | 78 | 49
Participants | 5 | 2
Statistical Analysis 1: Comparison: Arm A: G/P 300 mg/120 mg QD for 12 Wks vs Arm B: G/P 300 mg/120 mg QD for 16 Wks; Test type: Other — The difference in the percentage of subjects with post-treatment relapse between Arms A and B are summarized with two-sided 95% Wilson score intervals; Mean Difference (Final Values) = -2.50, 95% CI 2-sided [-10.49 to 5.49]

6. Secondary Outcome: Difference in On-Treatment Virologic Failure Between Arms C and D in Cirrhotic Subjects
Description: Difference in percentage of cirrhotic subjects experiencing on-treatment virologic failure (confirmed increase of > 1 log10 IU/mL above nadir during treatment, confirmed HCV RNA ≥ 100 IU/mL after HCV RNA < 15 IU/mL during treatment, or HCV RNA ≥ LLOQ at the end of treatment with at least 6 weeks of treatment) after 12 weeks of G/P with or without RBV for 12 weeks versus 16 weeks of G/P
Time Frame: Up to 28 weeks
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Groups:
- Arm D: G/P 300 mg/120 mg QD for 16 Wks: Cirrhotic subjects receiving Glecaprevir/Pibrentasvir (G/P) 300mg/120mg once daily for 16 weeks (G/P 300 mg/120mg QD for 16 Wks)
  Glecaprevir/Pibrentasvir (G/P) 300mg/120mg: daily
Arm/Group | Arm C: G/P 300 mg/120 mg QD + RBV 12 Wks | Arm D: G/P 300 mg/120 mg QD for 16 Wks
Number analyzed (Participants) | 21 | 29
Participants | 2 | 0
Statistical Analysis 1: Comparison: Arm C: G/P 300 mg/120 mg QD + RBV 12 Wks vs Arm D: G/P 300 mg/120 mg QD for 16 Wks; Test type: Other — Difference in percentage of subjects with on-treatment virologic failure between Arms C and D will be summarized with two-sided 95% Wilson score intervals; Mean Difference (Final Values) = 9.52, 95% CI 2-sided [-3.03 to 22.08]

7. Secondary Outcome: Difference in % of Relapse Between Cirrhotic Arms C & D
Description: Difference in the percentage of compensated cirrhotic subjects with post-treatment relapse (defined as confirmed HCV RNA>=Lower limit of quantification (LLOQ) between end of treatment and 12 weeks after last dose of study drug among subjects who completed treatment as planned with HCV RNA<LLOQ at end of treatment) after receiving 12 weeks G/P +/-Ribavirin (RBV) (Arm C) versus 16 weeks G/P (Arm D)
Time Frame: Up to 28 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm C: G/P 300 mg/120 mg QD + RBV 12 Wks | Arm D: G/P 300 mg/120 mg QD for 16 Wks
Number analyzed (Participants) | 21 | 20
Participants | 1 | 1
Statistical Analysis 1: Comparison: Arm C: G/P 300 mg/120 mg QD + RBV 12 Wks vs Arm D: G/P 300 mg/120 mg QD for 16 Wks; Excludes re-infection and death; Test type: Other; Mean Difference (Final Values) = -1.81, 95% CI 2-sided [-13.85 to 10.22]

8. Secondary Outcome: Difference in SVR12 Rates for 12-wk vs 16 wk
Description: Difference in proportions of SVR 12 rates will be determined for 12-week vs. 16-week treatment durations using contrasts within a logistic regression model with cirrhosis status and HCV genotype (1b vs non-1b) as factors
Time Frame: 28 weeks
Population: Modified Intent to Treat Population (mITT) analysis (All subjects enroll in Main study receiving at least one dose of study drug and according to the treatment arm in which they were actually treated)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: G/P 300 mg/120 mg QD for 12 Wks | Arm B: G/P 300 mg/120 mg QD for 16 Wks | Arm C: G/P 300 mg/120 mg QD + RBV 12 Wks | Arm D: G/P 300 mg/120 mg QD for 16 Wks
Number analyzed (Participants) | 78 | 49 | 21 | 29
Participants | 70 | 46 | 18 | 28
Statistical Analysis 1: Comparison: Arm A: G/P 300 mg/120 mg QD for 12 Wks vs Arm B: G/P 300 mg/120 mg QD for 16 Wks vs Arm C: G/P 300 mg/120 mg QD + RBV 12 Wks vs Arm D: G/P 300 mg/120 mg QD for 16 Wks; Test type: Other — Study was not powered to compare efficacy; p = 0.161, Chi-squared; Logistic regression contrast estimates with Wald confidence intervals and Chi-square p values; Logistic Regression Contrast Estimate = -0.812, 95% CI 2-sided [-1.947 to 0.323] — Comparison of Arm Pair A/C versus B/D overall on mITT population
Statistical Analysis 2: Comparison: Arm A: G/P 300 mg/120 mg QD for 12 Wks vs Arm B: G/P 300 mg/120 mg QD for 16 Wks vs Arm C: G/P 300 mg/120 mg QD + RBV 12 Wks vs Arm D: G/P 300 mg/120 mg QD for 16 Wks; Test type: Other — Study is not powered to compare efficacy of 12 wks vs 16 weeks of treatment; p = 0.890, Chi-squared; Logistic regression contrast estimates with Wald confidence intervals and Chi-square p values; Logistic regression contrast estimate = 0.890, 95% CI 2-sided [-1.239 to 1.076] — Difference in proportion of SVR12 rates for 12 vs 16 weeks on mITT Comparing Cirrhotic subjects versus non-cirrhotic subjects
Statistical Analysis 3: Comparison: Arm A: G/P 300 mg/120 mg QD for 12 Wks vs Arm B: G/P 300 mg/120 mg QD for 16 Wks vs Arm C: G/P 300 mg/120 mg QD + RBV 12 Wks vs Arm D: G/P 300 mg/120 mg QD for 16 Wks; Comparison of 12 weeks vs 16 weeks in Genotype 1b vs non-1b; Test type: Other — Study is not powered; p = 0.265, Chi-squared; Logistic regression contrast estimate = 0.977, 95% CI 2-sided [-0.740 to 2.694]

ADVERSE EVENTS:
Time Frame: 142 days
Arm/Group | Arm A: G/P 300 mg/120 mg QD for 12 Wks | Arm B: G/P 300 mg/120 mg QD for 16 Wks | Arm C: G/P 300 mg/120 mg QD + RBV 12 Wks | Arm D: G/P 300 mg/120 mg QD for 16 Wks
All-Cause Mortality (participants affected / at risk) | 1/78 | 0/49 | 0/21 | 0/29
Serious Adverse Events (participants affected / at risk) | 4/78 | 2/49 | 1/21 | 0/29
Other Adverse Events (participants affected / at risk) | 50/78 | 32/49 | 17/21 | 17/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: G/P 300 mg/120 mg QD for 12 Wks (N=78) | Arm B: G/P 300 mg/120 mg QD for 16 Wks (N=49) | Arm C: G/P 300 mg/120 mg QD + RBV 12 Wks (N=21) | Arm D: G/P 300 mg/120 mg QD for 16 Wks (N=29)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic Obstruction Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HCC final outcome Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Death related to HCC
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: G/P 300 mg/120 mg QD for 12 Wks (N=78) | Arm B: G/P 300 mg/120 mg QD for 16 Wks (N=49) | Arm C: G/P 300 mg/120 mg QD + RBV 12 Wks (N=21) | Arm D: G/P 300 mg/120 mg QD for 16 Wks (N=29)
Upper Respiratory Tract Infection (Infections and infestations) | 5 (5) | 0 (0) | 3 (3) | 2 (2)
Arthralgia (General disorders) | 4 (4) | 3 (3) | 2 (2) | 2 (2)
Fatigue (General disorders) | 13 (13) | 10 (10) | 10 (10) | 8 (8)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (7) | 7 (7) | 2 (2) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4) | 2 (2) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 15 (17) | 9 (9) | 7 (7) | 6 (7)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
This study did not include a group that received 16 weeks of glecaprevir and pibrentasvir with ribavirin.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/75/NCT03092375/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-08): https://cdn.clinicaltrials.gov/large-docs/75/NCT03092375/SAP_001.pdf